CLINICAL TRIAL: NCT03828110
Title: Investigating the Effectiveness of Robotic-Assisted Gait Training (RAGT) in the Rehabilitation of Children With Neurological Impairment Due to Acquired Brain Injury or Cerebral Palsy
Brief Title: The Effectiveness of Robotic Gait Training in Children With Neurological Impairment
Status: Completed | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: GIP-454
Record Dates: First submitted 2019-01-25; First posted 2019-02-04 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Acquired Brain Injury; Cerebral Palsy
Keywords: Robotic-Assisted Gait Training; Gait Rehabilitation
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with neurological impairment
  Interventions: Device: Robotic Assisted Gait Training (Lokomat); Procedure: Physiotherapy

INTERVENTIONS:
Device: Robotic Assisted Gait Training (Lokomat) — The RAGT treatment consisted of sessions lasting 45 minutes each performed with the commercially available Lokomat device. The same exercises were offered to the children with preset duration, speed, and difficulty. For all patients, the initial body-weight support was set at 50%, and was then gradually decreased according to the individual functional capacity. The guidance force was initially set to 100% for all children, and then gradually reduced.
  Other Names: RAGT
Procedure: Physiotherapy — The physiotherapic sessions aimed at strengthening the gluteus and quadriceps muscles, stretching the hip flexor and hamstrings muscles, increasing static balance, increasing dynamic balance, increasing functional abilities, improving ground gait and climbing stairs.

SUMMARY:
The recovery of walking ability is one of the primary rehabilitation goals for children with neurological impairment. The aim of the study is to investigate the clinical effectiveness of rehabilitation treatments based of Robotic-Assisted Gait Training (RAGT). Additional goals of the research are to identify the specific effects of RAGT in children with different etiologies (acquired brain injury and cerebral palsy) and with different levels of function (according to the Gross Motor Function Classification System).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acquired brain injury in pediatric age and adolescence (4 to 18 years) or cerebral palsy;
* Femur length of at least 23 cm;
* Patients able to signal pain, fear or discomfort reliably and to follow simple instructions.

Exclusion Criteria:

* injection of botulinum toxin during the 6 months prior to the enrollment;
* oral medications reducing muscle tone;
* previous orthopedic surgery;
* severe lower-extremity contractures;
* fractures or osseous instabilities;
* osteoporosis;
* contraindication of full body load due to previous surgeries;
* severe retarded bone growth;
* unhealed skin lesions in the lower-extremities;
* thromboembolic diseases
* cardiovascular instability
* acute or progressive neurological disorders
* aggressive or self-harming behavior.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Neurophysiatric care unit
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in 6minWT distance walked | After four weeks of treatment
  The 6-minute walk test (6minWT) was used to assess endurance during self-paced, submaximal walk by measuring the distance walked within 6 minutes along a standardized route through the hospital corridors.
change in GMFM-88: total score and Dimensions | After four weeks of treatment
  The Gross Motor Function Measure (GMFM) measures the child's overall functional abilities, and is divided into the following sections: (A) lying and rolling, (B) sitting, (C) crawling and kneeling, (D) standing, and (E) walking, running, and jumping.

SECONDARY OUTCOMES:
change in spatiotemporal gait parameters | After four weeks of treatment
  Data obtained using 3D gait analysis
change in kinematic gait parameters | After four weeks of treatment
  Data obtained using 3D gait analysis
change in kinetic gait parameters | After four weeks of treatment
  Data obtained using 3D gait analysis
change in FAQ score | After four weeks of treatment
  The Functional Activities Questionnaire (FAQ) measures instrumental activities of daily living
Lokomat therapy duration | After four weeks of treatment
  Total duration of therapy sessions (hours and minutes)
Lokomat therapy total distance walked | After four weeks of treatment
  Total distance walked during sessions (in meters)
Lokomat therapy total time walked | After four weeks of treatment
  Total time walked during sessions
Lokomat stiffness values (LStiff) | After four weeks of treatment
  Joint stiffness measured by the Lokomat device (in Newton/meters)
Lokomat force values (LForce) | After four weeks of treatment
  Joint force measured by the Lokomat device (in Newton)

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Biffi, PhD, Principal Investigator — Scientific Institute IRCCS "E. Medea"
Locations (1):
- Scientific Institute IRCCS E. Medea, Bosisio Parini, Lecco, Italy

REFERENCES:
- [Derived] Beretta E, Storm FA, Strazzer S, Frascarelli F, Petrarca M, Colazza A, Cordone G, Biffi E, Morganti R, Maghini C, Piccinini L, Reni G, Castelli E. Effect of Robot-Assisted Gait Training in a Large Population of Children With Motor Impairment Due to Cerebral Palsy or Acquired Brain Injury. Arch Phys Med Rehabil. 2020 Jan;101(1):106-112. doi: 10.1016/j.apmr.2019.08.479. Epub 2019 Sep 25. PMID 31562873